CLINICAL TRIAL: NCT04086875
Title: A Mobile TXT-Based Intervention to Improve Adherence to Adjuvant Hormone Therapy and Symptom Management for BCa Survivors
Brief Title: A Text-based Intervention in Improving Adherence to Hormone Therapy in Patients With Stage I-III Hormone Receptor Positive Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kuang-Yi Wen, Associate Professor - Medical Oncology, Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19F.265; R01CA222246 (NIH)
Record Dates: First submitted 2019-09-04; First posted 2019-09-12 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Estrogen Receptor Positive Tumor; Progesterone Receptor Positive Tumor; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8
MeSH Terms: interventions — Focus Groups; Communication Devices for People with Disabilities; Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase 1 (focus groups) (Experimental): Participants attend focus groups on adherence to hormone therapy.
  Interventions: Behavioral: Focus Group; Other: Questionnaire Administration
- Phase II Group 1 (text messages) (Experimental): Participants receive text messages twice weekly for 6 months to remind and motivate participants about AHT adherence.
  Interventions: Other: Text Message; Other: Questionnaire Administration
- Phase II Group II (usual care) (Active Comparator): Participants receive usual care.
  Interventions: Other: Best Practice; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Focus Group — Participate in focus group
  Arms: Phase 1 (focus groups)
Other: Text Message — Receive text messages
  Other Names: SMS Text; SMS Text Message; Text
  Arms: Phase II Group 1 (text messages)
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
  Arms: Phase II Group II (usual care)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies how well a text-based intervention works in improving adherence to hormone therapy in patients with stage I-III hormone receptor positive breast cancer. Women often require long term therapy with adjuvant hormone therapy to prevent the cancer from returning and to improve overall survival. Side effects from hormone therapy may prevent some women from staying adherent to their medication therapy. A text-based intervention may provide educational information to breast cancer patients who are undergoing adjuvant hormone therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Examine the efficacy of messaging for adjuvant hormone therapy compliance promotion (mAHT-CaP) in a randomized control trial (RCT) design.

SECONDARY OBJECTIVES:

I. Conduct mediator analyses of intervention efficacy..

EXPLORATORY OBJECTIVES:

I. Explore whether age (=< 45 versus [vs.] > 45 at diagnosis) and race/ethnicity (white vs. non-white) moderate intervention effects on medication adherence and symptom distress.

OUTLINE:

PHASE I: Participants attend focus groups on adherence to hormone therapy.

PHASE II: Participants are randomized to 1 of 2 groups.

GROUP I: Participants receive text messages twice weekly for 6 months to remind and motivate participants about adjuvant hormonal therapy (AHT) adherence.

GROUP II: Participants receive usual care.

After completion of study, participants are followed up at 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Woman diagnosed with stage I-III breast cancer (BCa).
* Hormone receptor positive tumor.
* Completed local definitive treatment (i.e., surgery chemotherapy, radiation).
* Within 3 month of initiation of a new adjuvant hormonal therapy (AHT) regimen.
* At least 12 months of AHT recommended.
* Able to read and understand English.
* Able to provide informed consent.
* Have a mobile device with text (TXT) capability.
* Know or willing to learn how to use TXT.

Exclusion Criteria:

• Cognitive impairment documented in the electronic medical record (EMR), biological variables (sex).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2024-09-24 (Estimated); Study Completion 2024-09-24 (Estimated)

PRIMARY OUTCOMES:
Adjuvant hormone therapy (AHT) adherence | Up to 12 months
  Assessed by wireless smart pill bottles for all participants. Daily adherence will be defined as accessing the pill bottle once per 24 hour period. Proportion adherence will be summarized by week and study arm, and presented graphically.
Symptom distress | Up to 12 months
  Measured by the Breast Cancer Prevention Trial Symptom Scale, which has sound psychometric properties in breast cancer (BCa) patients. There are a total of 43 items in the scale across eight domains. Each item is a five-point Likert scale, ranging from 0 (not at all) to 4 (extremely), used to rate symptoms. Items accounting for side effects specifically related to AHT (e.g., bone pain) and other general symptoms (e.g., constipation) are added. Participants are asked whether they are bothered by each symptom and whether they think it related to their AHT or not. The two resulting scales consist of the sum of the endorsed symptom total each woman does or does not attribute to AHT.

SECONDARY OUTCOMES:
Cognitive-affective barriers for AHT adherence | Up to 12 months
  Will be developed and will test the mediating effect of cognitive affective barriers on proportion of days adherent (average over 12 months)
Cognitive-affective barriers for symptom distress | Up to 12 months
  Will be developed and will test the mediating effect of cognitive affective barriers on the difference between baseline and 12-month symptom distress. Symptom distress is measured by the Breast Cancer Prevention Trial Symptom Scale

OTHER OUTCOMES:
Perceived benefits | Up to 12 months
  Measured by the Health Beliefs and Medication Adherence in Breast Cancer.
Perceived susceptibility | Up to 12 months
  Measured by the Health Beliefs and Medication Adherence in Breast Cancer.
Knowledge and self-efficacy for taking AHT | Up to 12 months
  Measured by the Medication Understanding and Use Self-Efficacy Scale. This scale is a total of 8 questions with a total score ranging from 0 to 24. It measures patients' self-efficacy in understanding and using medication.
Self-efficacy for managing symptoms: modified version of Lorig's Chronic Disease Self-Efficacy Scale | Up to 12 months
  Measured by a modified version of Lorig's Chronic Disease Self-Efficacy Scale for managing symptoms. The modified scale asks participants concerning their certainty of controlling symptoms caused by AHT in order to perform daily activities. The scale is a 6 item questionnaire on a 10-point Likert scale. Score is the mean of the six items, with higher scores indicating higher self-efficacy.
Affective distress about AHT | Up to 12 months
  Assessed by The Intrusion subscale of the Revised Impact of Events Scale, a well validated instrument that measures stress-related intrusive thoughts. The Intrusion subscale consists of 8 items with scores for each item ranging from 0 to 4.
Social support | Up to 12 months
  Measured using the Multidimensional Scale of Perceived Social Support (MSPSS). The MSPSS assesses perceptions of support received from family, friends, and significant others, which reflect distinct reliable and valid factors in BCa patient samples and medication adherence studies. This scale consists of 12 items on a 7-point Likert scale (1 very strongly disagree, 7 very strongly agree). Total score is calculated by adding the score across all items and dividing by 12. Scores of 5.1-7 are high social support.

CONTACTS AND LOCATIONS:
Overall Officials: Kuang-Yi Wen, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (7):
- United States (7):
  - Jefferson Health - South Jersey, Sewell, New Jersey
  - Jefferson Health - Abington, Abington, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Jefferson Health - Northeast (Aria Torresdale), Philadelphia, Pennsylvania
  - Thomas Jefferson University - Methodist Hospital, Philadelphia, Pennsylvania